CLINICAL TRIAL: NCT00993668
Title: A Phase 4, Randomized, Single-blind, Placebo-controlled, Multicenter Study to Evaluate the Immunogenicity of Pneumococcal and Influenza Vaccines in Adult Subjects With Rheumatoid Arthritis Receiving Certolizumab Pegol or Placebo
Brief Title: Assessing the Use of Certolizumab Pegol in Adult Subjects With Rheumatoid Arthritis on the Antibody Response When Receiving Influenza Virus and Pneumococcal Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RA0017
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Results first posted 2011-06-20 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2012-01

CONDITIONS: Rheumatoid Arthritis
Keywords: influenza; vaccine; pneumococcal vaccine; certolizumab pegol; Cimzia
MeSH Terms: conditions — Arthritis, Rheumatoid; Influenza, Human | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- Cimzia (Experimental): Certolizumab pegol
  Interventions: Biological: Certolizumab pegol

INTERVENTIONS:
Other: Placebo — Placebo - Two 0.9% saline subcutaneous (sc) injections at Week 0, Week 2, and Week 4 followed by two sc injections of Open-Label (OL) CZP 200 mg at Weeks 6, 8 and 10, then one sc injection of OL CZP 200 mg every two weeks from Week 12 until last drug administration (up to Week 32).
  Arms: Placebo
Biological: Certolizumab pegol — Certolizumab pegol - Two 200 mg subcutaneous (sc) injections at Week 0, Week 2, and Week 4 followed by one sc injection of Open-Label (OL) CZP 200 mg from Week 6 until last drug administration (up to Week 32).
  Other Names: Cimzia®
  Arms: Cimzia

SUMMARY:
The purpose of this trial is to assess the affect of Certolizumab Pegol (CZP) treatment on antibody response to T cell-independent and T cell-dependent immunizations using pneumococcal and influenza vaccines, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years old at the screening visit
* Subjects must be able to understand the information provided to them and to give written informed consent, and be able and willing to comply with the study requirements
* Female subjects must be either postmenopausal for at least 1 year, surgically incapable of childbearing, or effectively practicing an acceptable method of contraception (either oral/parenteral/implantable hormonal contraceptives, intrauterine device or barrier and spermicide. Abstinence only is not an acceptable method. Subjects must agree to use adequate contraception during the study and for 10 weeks after the last dose of CZP. Male subjects must agree to ensure they or their female partner(s) use adequate contraception during the study and for 10 weeks after the subject receives their last dose of CZP
* Subjects must have a diagnosis of adult-onset Rheumatoid Arthritis (RA) of at least 6-months duration as defined by the 1987 American College of Rheumatology (ACR) classification criteria
* Subjects must have active RA disease as defined by: ≥ 4 tender joints (28 joint count) at Screening and Week 0; and ≥ 4 swollen joints (28 joint count) at Screening and Week 0

Exclusion Criteria:

* Subjects who have a diagnosis of any other inflammatory arthritis (eg., psoriatic arthritis or ankylosing spondylitis)
* Subjects who have a history of an infected joint prosthesis at any time with that prosthesis still in situ
* Subjects must be free of defined prohibited medication and biological therapy
* Subjects who have received any experimental nonbiological therapy, within or outside of a clinical trial in the 3 months prior to Week 0
* Subjects who have received any experimental biological agent in the past 3 months or within 5 half-lives prior to Week 0 (whichever is longer)
* Subjects who have received previous treatment with biological response modifier therapy for RA that resulted in a severe hypersensitivity reaction or an anaphylactic reaction.
* Subjects with a history of pneumococcal or influenza infection in the last 3 months
* Subjects with a history of pneumococcal vaccination in the last 5 years
* Subjects with a history of influenza vaccination within the last 6 months
* Female subjects who are breast-feeding, pregnant, or plan to become pregnant during the trial or within 3 months following last dose of study drug
* Subjects with a history of chronic or recurrent infections (more than 3 episodes requiring antibiotics/antivirals during the preceding year), recent serious or life-threatening infection within 6 months (including herpes zoster), or any current sign or symptom that may indicate an infection
* Subjects who have had a splenectomy
* Subjects who have had a hypersensitivity reaction to previous pneumococcal or influenza vaccination
* Subjects who have a known hypersensitivity to eggs and egg products or to other components of the vaccine
* Subjects with a history of Guillain-Barre syndrome
* Subjects with a history of tuberculosis, active tuberculosis, positive chest x-ray for tuberculosis, or positive purified protein derivative (PPD) skin test (defined as induration of ≥5 mm). Subjects who are not candidates for PPD testing due to prior severe reaction to the PPD test or a history of PPD positivity must undergo an Elispot test instead for tuberculosis evaluation. Subjects testing positive via the PPD or having an indeterminate or positive Elispot test, or for which latent tuberculosis cannot be ruled out, may be enrolled in the study provided that they are treated (eg., isoniazid for 9 months) and that their treatment has been initiated at least 4 weeks prior to the first administration of CZP
* Subjects at high risk of infection (eg., presence of leg ulcers or an indwelling urinary catheter, persistent or recurrent chest infections, bedridden or wheelchair bound subjects)
* Subjects with a history of a lymphoproliferative disorder including lymphoma or signs and symptoms suggestive of lymphoproliferative disease
* Subjects with known concurrent acute or chronic viral hepatitis B or C or positive hepatitis B surface antigen (HBs-Ag) or hepatitis C virus antibody (HCV-Ab)
* Subjects with known human immunodeficiency virus (HIV) infection
* Subjects receiving any live or attenuated vaccination within 12 weeks prior to Week 0
* Concurrent malignancy or a history of malignancy (other than carcinoma of the cervix or basal cell carcinoma successfully treated more than 5 years prior to screening)
* Subjects with Class III or Class IV congestive heart failure according to the New York Heart Association (NYHA) 1964 classification criteria
* Subjects with a history of, or suspected, demyelinating disease of the central nervous system (eg., multiple sclerosis or optic neuritis)
* Subjects with a current or recent history of severe, progressive, and/or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological or cerebral disease
* Subjects with any other condition (eg., clinically significant laboratory values) which in the Investigator's judgement would make the subject unsuitable for inclusion in the study
* Subjects with a history of an adverse reaction to polyethylene glycol (PEG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1-877-822-9493 (UCB)
Locations (41):
- United States (41):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Tuscaloosa, Alabama
  - Peoria, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Los Angeles, California
  - Palm Desert, California
  - Santa Maria, California
  - Santa Monica, California
  - Aventura, Florida
  - Fort Lauderdale, Florida
  - Melbourne, Florida
  - Orange Park, Florida
  - Palm Harbor, Florida
  - Venice, Florida
  - Vero Beach, Florida
  - Zephyrhills, Florida
  - Idaho Falls, Idaho
  - Meridian, Idaho
  - Cedar Rapids, Iowa
  - Kalamazoo, Michigan
  - Lansing, Michigan
  - Hattiesburg, Mississippi
  - Florissant, Missouri
  - Reno, Nevada
  - Brooklyn, New York
  - Smithtown, New York
  - Syracuse, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Middleburg Heights, Ohio
  - Oklahoma City, Oklahoma
  - Duncansville, Pennsylvania
  - Erie, Pennsylvania
  - West Reading, Pennsylvania
  - Myrtle Beach, South Carolina
  - Orangeburg, South Carolina
  - San Antonio, Texas
  - Seattle, Washington
  - Oak Creek, Wisconsin

REFERENCES:
- [Derived] Kivitz AJ, Schechtman J, Texter M, Fichtner A, de Longueville M, Chartash EK. Vaccine responses in patients with rheumatoid arthritis treated with certolizumab pegol: results from a single-blind randomized phase IV trial. J Rheumatol. 2014 Apr;41(4):648-57. doi: 10.3899/jrheum.130945. Epub 2014 Mar 1. PMID 24584918
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started in September of 2009 with recruitment occurring in the United States. The primary outcome completed in June 2010 and the open-label extension completed in February 2011.
Pre-assignment Details: Treatment column headings reflect the treatment received in the Single-Blind (SB) period.
Groups:
- Cimzia: Certolizumab pegol - Two 200 mg subcutaneous (sc) injections at Week 0, Week 2, and Week 4 followed by one sc injection of Open-Label (OL) CZP 200 mg from Week 6 until last drug administration (up to Week 32).
Period: Single-Blind Period
Arm/Group | Placebo | Cimzia
Started | 114 | 110
Completed | 110 | 107
Not Completed | 4 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 3 | 1
Period: Open-Label Period
Arm/Group | Placebo | Cimzia
Started | 109 (1 subject chose not to enter the optional open-label period) | 106 (1 subject chose not to enter the optional open-label period)
Completed | 86 | 91
Not Completed | 23 | 15
Not completed — Adverse Event | 9 | 8
Not completed — Lack of Efficacy | 4 | 3
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cimzia | Total
Number analyzed (Participants) | 114 | 110 | 224
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 102 | 94 | 196
  >=65 years | 12 | 16 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.65 (11.12) | 53.05 (11.78) | 52.85 (11.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 92 | 179
  Male | 27 | 18 | 45
Region of Enrollment [Number; unit: participants]
  United States | 114 | 110 | 224

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Without Baseline Protective Titers Achieving a ≥ 2-fold Titer Increase in ≥ 3 of 6 Pneumococcal Antigens (6B, 9V, 14, 18C, 19F, and 23F) at Week 6.
Time Frame: Baseline, End of single blind period (Week 6)
Population: Of the 224 randomized subjects (114 Placebo, 110 CZP), 176 were in the Per Protocol Set Pneumococcal (PPSP) population (88 Placebo, 88 CZP) without baseline protective titers, and are included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cimzia
Number analyzed (Participants) | 88 | 88
percentage of participants | 62.5 [52.4 to 72.6] | 54.5 [44.1 to 64.9]

2. Primary Outcome: Percentage of Subjects Without Baseline Protective Titers Achieving a ≥ 4-fold Titer Increase in ≥ 2 of 3 Influenza Antigens (2009/2010 Composition) at Week 6.
Time Frame: Baseline, End of single blind period (Week 6)
Population: Of the 224 randomized subjects (114 Placebo, 110 CZP), 169 were in the Per Protocol Set Influenza (PPSI) population (83 Placebo, 86 CZP) without baseline protective titers, and are included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cimzia
Number analyzed (Participants) | 83 | 86
percentage of participants | 61.4 [51.0 to 71.9] | 53.5 [42.9 to 64.0]

3. Secondary Outcome: Percentage of All Subjects Achieving a ≥ 2-fold Titer Increase in ≥ 3 of 6 Pneumococcal Antigens (6B, 9V, 14, 18C, 19F, and 23F) at Week 6.
Time Frame: End of single blind period (Week 6)
Population: Of the 224 randomized subjects (114 Placebo, 110 CZP), 217 were in the Full Analysis Set Pneumococcal (FASP) population (110 Placebo, 107 CZP), and are included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cimzia
Number analyzed (Participants) | 110 | 107
percentage of participants | 58.2 [49.0 to 67.4] | 53.3 [43.8 to 62.7]

4. Secondary Outcome: Percentage of All Subjects Achieving a ≥ 4-fold Titer Increase in ≥ 2 of 3 Influenza Antigens (2009/2010 Composition) at Week 6.
Time Frame: End of single blind period (Week 6)
Population: Of the 224 randomized subjects (114 Placebo, 110 CZP), 109 were in the Full Analysis Set Influenza (FASI) population (109 Placebo, 107 CZP), and are included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cimzia
Number analyzed (Participants) | 109 | 107
percentage of participants | 54.1 [44.8 to 63.5] | 50.5 [41.0 to 59.9]

5. Secondary Outcome: Percentage of Subjects With no Previous Protective Pneumococcal Antibody Titers at Baseline With Protective Pneumococcal Antibody Titers (≥1.6 µg/ml in ≥ 3 of 6 of the Pneumococcal Antigens) at Week 6.
Time Frame: Baseline, End of single blind period (Week 6)
Population: Of the 224 randomized subjects (114 Placebo, 110 CZP), 180 were in the Per Protocol Set Pneumococcal (PPSP) population (90 Placebo, 90 CZP) without baseline protective titers. Of these 180 subjects 150 (75 Placebo, 75 CZP) had protective pneumococcal antibody titers and are included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cimzia
Number analyzed (Participants) | 75 | 75
percentage of participants | 57.3 [46.1 to 68.5] | 50.7 [39.4 to 62.0]

6. Secondary Outcome: Percentage of Subjects With no Previous Protective Influenza Antibody Titers at Baseline With Protective Influenza Antibody Titers (≥1:40 in ≥ 2 of 3 Influenza Antigens) at Week 6.
Time Frame: Baseline, End of single blind period (week 6)
Population: Of the 224 randomized subjects (114 Placebo, 110 CZP), 169 were in the Per Protocol Set Influenza (PPSI) population (83 Placebo, 86 CZP) without baseline protective titers but with protective influenza antibody titers, and are included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cimzia
Number analyzed (Participants) | 83 | 86
percentage of participants | 73.5 [64.0 to 83.0] | 64.0 [53.8 to 74.1]

7. Secondary Outcome: Percentage of All Subjects With Protective Pneumococcal Antibody Titers (≥1.6 µg/ml in ≥ 3 of 6 of the Pneumococcal Antigens) at Week 6.
Time Frame: End of single blind period (Week 6)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cimzia
Number analyzed (Participants) | 110 | 107
percentage of participants | 65.5 [56.6 to 74.3] | 62.6 [53.4 to 71.8]

8. Secondary Outcome: Percentage of All Subjects With Protective Influenza Antibody Titers (≥1:40 in ≥ 2 of 3 Influenza Antigens) at Week 6.
Time Frame: End of single blind period (Week 6)
Population: Of the 224 randomized subjects (114 Placebo, 110 CZP), 216 were in the Full Analysis Set Influenza (FASI) population (109 Placebo, 107 CZP), and are included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cimzia
Number analyzed (Participants) | 109 | 107
percentage of participants | 77.1 [69.2 to 85.0] | 71.0 [62.4 to 79.6]

9. Secondary Outcome: Percentage of Subjects Without Baseline Protective Titers Achieving a ≥ 2-fold Titer Increase in ≥ 3 of 6 Pneumococcal Antigens at Week 6 by Concomitant Methotrexate (MTX) Use.
Time Frame: Baseline, End of single blind period (Week 6)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cimzia
Number analyzed (Participants) | 88 | 88
percentage of participants
  Concomitant MTX Use (n=60, 63) | 50.0 [37.3 to 62.7] | 44.4 [32.2 to 56.7]
  No Concomitant MTX Use (n=28, 25) | 89.3 [77.8 to 100.00] | 80.0 [64.3 to 95.7]

10. Secondary Outcome: Percentage of Subjects Without Baseline Protective Titers Achieving a ≥ 4-fold Titer Increase in ≥ 2 of 3 Influenza Antigens at Week 6 by Concomitant MTX Use.
Time Frame: Baseline, End of single blind period (Week 6)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cimzia
Number analyzed (Participants) | 83 | 86
percentage of participants
  Concomitant MTX Use (n=57, 59) | 50.9 [37.9 to 63.9] | 45.8 [33.1 to 58.5]
  No Concomitant MTX Use (n=26, 27) | 84.6 [70.7 to 98.5] | 70.4 [53.1 to 87.6]

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) data summarized in the first two columns refer to the 6-week Single-Blind (SB) period of the study. The final column refers to AE data collected on subjects who received Cimzia at any time during the study (up to 42 weeks).
Groups:
- Placebo (Single Blind): Placebo - Two 0.9% saline subcutaneous injections at Week 0, Week 2, and Week 4
- Cimzia (Single Blind): Certolizumab pegol - Two 200 mg subcutaneous injections at Week 0, Week 2, and Week 4
- Cimzia at Any Time: Certolizumab pegol (at any time) - Subjects randomized to receive Certolizumab pegol (CZP) during the single blind (SB) period will receive two subcutaneous (sc) injections of SB CZP 200 mg at Weeks 0, 2, and 4 followed by one sc injection of Open-Label (OL) CZP 200 mg from Week 6 until last drug administration (up to Week 32). Subjects randomized to placebo during the SB period will receive two 0.9% saline sc injections at Week 0, Week 2, and Week 4, followed by two sc injections of OL CZP 200 mg at Weeks 6, 8 and 10, then one sc injection of CZP 200 mg every two weeks from Week 12 until last drug administration (up to Week 32).
Arm/Group | Placebo (Single Blind) | Cimzia (Single Blind) | Cimzia at Any Time
Serious Adverse Events (participants affected / at risk) | 1/114 | 2/110 | 15/219
Other Adverse Events (participants affected / at risk) | 29/114 | 22/110 | 155/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Single Blind) (N=114) | Cimzia (Single Blind) (N=110) | Cimzia at Any Time (N=219)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 4 (5)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Latent Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Chest Wall Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Chordoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Depressed Level Of Consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Granuloma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Single Blind) (N=114) | Cimzia (Single Blind) (N=110) | Cimzia at Any Time (N=219)
Nausea (Gastrointestinal disorders) | 6 (6) | 6 (7) | 20 (22)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 2 (2) | 18 (22)
Fatigue (General disorders) | 5 (5) | 2 (2) | 18 (20)
Pain (General disorders) | 4 (7) | 4 (4) | 11 (15)
Nasopharyngitis (Infections and infestations) | 6 (6) | 10 (10) | 31 (36)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (6) | 4 (4) | 30 (32)
Sinusitis (Infections and infestations) | 5 (5) | 2 (2) | 23 (28)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 4 (4) | 17 (17)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0) | 14 (16)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 16 (19)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 (6) | 0 (0) | 11 (18)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 20 (26)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (8) | 3 (3) | 15 (25)
Headache (Nervous system disorders) | 15 (23) | 8 (12) | 28 (71)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 13 (16)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 2 (2) | 23 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 18 (18)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 14 (15)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5) | 15 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.